CLINICAL TRIAL: NCT04919044
Title: Effect of Motor Imagery Training On Quadriceps Strength In Community Dwelling Elderly
Brief Title: Motor Imagery Training in Community Dwelling Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Principal Investigator, Imtiyaz Ali Mir, Principal Investigator, Universiti Tunku Abdul Rahman
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UMFD3026-4
Record Dates: First submitted 2021-06-02; First posted 2021-06-09 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Old Age; Debility
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor did not know participants belonged to which group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Imagery (Experimental): The participants were instructed to imagine and visualize to straighten both knees with eyes closed. You have to see and feel only what you would see and feel if you had to perform the action to straighten both of your knees in sitting position. Imagine the movement using the most comfortable way for you, and make sure not to contract your muscles.
  Interventions: Other: Motor Imagery Training
- Control (No Intervention): No intervention provided.

INTERVENTIONS:
Other: Motor Imagery Training — The number of imagined contractions were 34 trials, each trial was 10 seconds with 5seconds rest between each trial and 2 minutes' rest was given after first 17 trials.
  Arms: Motor Imagery

SUMMARY:
An aging society is known as having at least 7% of its population aged 65 and older, whereas 14% or more known to be an aged nation. Age has a detrimental effect on the physical performance and the muscle strength, the reduced muscle strength, mass and structure in the elderly are due to aging, disuse and inactivity. In the elderly, the reduction of muscle strength is faster than the associated loss of muscle mass. The maximum isometric strength of knee extensors and muscle mass decrease due to aging. The combination of quadriceps and handgrip strength weakness in the elderly is associated with the poorest scores on quality of life, GP contact-time, gait speed, hospitalization and disability in daily living. Quadriceps weakness among elderly is also proved to be a contributing factor to fall among frail nursing home residents. A systematic review and meta-analysis revealed that quadriceps muscle weakness was associated with greater risk of developing knee osteoarthritis during 2.5 to 14 year follow-up in either gender. In overall, aging cause reduce muscle strength, especially quadriceps muscle, can cause many others negative consequences, thus a study of effect motor imagery on quadriceps muscle strength in community-dwelling elderly should be carried out, if this study is proven to effectively, motor imagery technique can be widely utilized on bedridden elderly or elderly who have severe cardiovascular disease who unable to perform physical activity to maintain or improve their muscle strength.

DETAILED DESCRIPTION:
The decrease in the number of skeletal muscle and decline in muscle function is the most important factor in influencing the ability to perform physical function independently in the later stage of our life. The reduction of quadriceps strength with advancing age in both gender is proved to be associated with an increased risk of fractures, increased chance of worsening of knee pain, high risk of osteoarthritis. Quadriceps weakness is also proved to be a contributing factor to falls among frail nursing home residents.

Motor imagery had been widely utilized and proved to benefits different population. Motor imagery training makes a better motor performance as proved to be an effective tool in stroke rehabilitation, it is effective and useful when there are severely injured patients. This imagery training has turned into performance enrichment ways and simulation tools which has been widely utilized in sports psychological interventions as well.

Motor imagery can be defined as a dynamic mental state during which the representation of a given motor act or movement is rehearsed in working memory without any overt motor output. Motor imagery can also be defined as utilizing whole senses to reform or form an experience in one's thought. Motor imagery can be performed in different modes which can be classified into visual, tactile, auditory, gustatory, olfactory, and kinesthetic modes. There are lot of studies which have showed that motor imagery task does activate the cortical and subcortical regions of the brain and they overlap in a great extent with task required movement execution. The parts of the brain proved to participate in motor control consists of the premotor cortex (PMC), supplementary motor area (SMA), as well as the primary motor cortex (M1). All these brain areas are nearly related to the basal ganglia and cerebellum, as a result, large feedback loop systems are formed. The aim of this research is to investigate the effect of motor imagery training on quadriceps strength among community-dwelling elderly. The second aim of our study is to compare the gender differences with regards to quadriceps muscle improvement after motor imagery training.

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* Aged 60 and above
* Participant who has a mean score of more than 3 in Movement Imagery Questionnaire-3
* Participant who scored 22 and above in MONTREAL COGNITIVE ASSESSMENT (MOCA) VERSION 7.1

Exclusion Criteria:

* Individual with neurological impairment or musculoskeletal injury.
* Participants unable to follow the instructions.
* Individuals using any anti-epileptic drugs and/or psychiatric drugs.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-08-08 (Actual); Primary Completion 2022-02-10 (Estimated); Study Completion 2022-02-10 (Estimated)

PRIMARY OUTCOMES:
Quadriceps Strength | Change from baseline Quadriceps strength at 4 weeks
  The participants were in sitting position, hand-held dynamometer was place on the shin of the tibia just above medial and lateral malleolus. Before measuring the quadriceps strength, participant's knees were held in 90-degree flexion and feet not in contact with the floor. The participants were instructed to straighten leg by pushing against hand-held dynamometer. Peak force generated by dynamometer was recorded. The measurement was repeated three times to take an average of 3.

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Tunku Abdul Rahman, Kajang, Selangor, Malaysia